CLINICAL TRIAL: NCT05984134
Title: Efficacy and Safety of Recombinant Human Thymosin β4(NL005) for Injection in Patients With Acute Myocardial Infarction: a Phase IIb Clinical Study
Brief Title: Efficacy and Safety Study of Thymosin Beta 4 in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL005-AMI-IIb
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acute Myocardial Infarction
Keywords: CMR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Middle Dose (Experimental): 12 hours after PCI: 0.5 ug/kg Recombinant Human Thymosin β4 （intravenous injection），Day2-Day7 after PCI：0.5 ug/kg Recombinant Human Thymosin β4 （intravenous injection）
  Interventions: Drug: NL005 Middle Dose
- High Dose (Experimental): 12 hours after PCI: 1.0 ug/kg Recombinant Human Thymosin β4 （intravenous injection），Day2-Day7 after PCI：1.0 ug/kg Recombinant Human Thymosin β4 （intravenous injection）
  Interventions: Drug: NL005 High Dose
- Placebo (Placebo Comparator): Patients in this treatment group will receive placebo respective. Continuous administration for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NL005 Middle Dose — Patients in this treatment group will receive NL005 for 0.5 ug/kg respective.Continuous administration for 7 days.
  Other Names: NL005（ Middle Dose）
  Arms: Middle Dose
Drug: NL005 High Dose — Patients in this treatment group will receive NL005 for 1.5 ug/kg respective.Continuous administration for 7 days.
  Other Names: NL005（ High Dose）
  Arms: High Dose
Drug: Placebo — 30 subjects will be randomly assigned to the placebo for 7 days
  Arms: Placebo

SUMMARY:
A multicenter randomized double-blind placebo parallel control design was used in this study. The 90 participants were randomly assigned to placebo, 0.5μg/kg dose group, and 1.0μg/kg dose group in a ratio of 1:1:1. After randomization, subjects received the trial drug or placebo intravenously within 12 hours and on days 2 to 7 after PCI. The patients were observed 90 days after PCI.

DETAILED DESCRIPTION:
Cardiovascular magnetic resonance imaging (CMR) was performed on day 5 and day 90 after PCI to evaluate myocardial infarction size, microvascular obstruction area, left ventricular ejection fraction (LVEF), left ventricular end-systolic volume (LVESV), and left ventricular end-diastolic volume (LVEDV). Physical examination, blood routine examination, and coagulation function examination were performed before the first dose, on the 7th, 30th, and 90th day after PCI. The examination before the first dose was conducted to accept the examination results from the current onset to the first dose.Electrocardiogram (ECG) was performed before the first dose, day 2, day 7, day 30, and day 90 after PCI, and the test results from the period after PCI to the first dose were received. Vital signs were examined before the first dose, day 1 to day 7, day 30, and day 90 after PCI, and the results of the examination from the first onset to the first dose were accepted during the examination before the first dose. Blood biochemical tests were performed before the first dose, from day 2 to day 4, day 7, day 30, and day 90 after PCI. The results of the examinations from the first onset to the first dose were accepted during the examination before the first dose. High-sensitivity troponin I(hs-cTnI) or troponin I(cTnI) and amino-terminal B-type natriuretic peptide precursor (NT-proBNP) or B-type natriuretic peptide (BNP) were tested before first administration and on days 2, 3, 4, and 7 after PCI. Examination results from the time after PCI to the time before initial administration; Creatine kinase isoenzyme (CK-MB) tests were performed before the first dose, 12 hours after the first dose, day 2 (if it coincided with 12 hours after the first dose, no repeat blood collection was required), day 3, and day 4. The test results from the period after PCI to the period before the first dose were accepted. Tumor markers were detected and immunogenic blood samples were collected before the first dose and on the 30th day after PCI. The tumor markers were examined before the first dose. Urine routine examination was performed before the first dose and on the 90th day after PCI. The examination before the first dose accepted the examination results from the onset of the disease to the first dose. Drug combinations, adverse events, and cardiovascular events were recorded during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects or their guardians voluntarily participate in the experiment and sign the informed consent;
2. Age ≥18 years old and ≤75 years old, gender is not limited;
3. STEMI patients with proximal or/and middle occlusion of a single left anterior descending artery (TIMI grade 0-1) and PCI;
4. No coronary collateral (Rentrop grade 0);
5. meet one of the following conditions:

   * The total myocardial ischemia time before PCI was < 6 hours, and the TIMI grade after PCI was < 3
   * 6 hours ≤ Total myocardial ischemia time before PCI ≤24 hours Note: Total myocardial ischemia time =PCI wire passage time - start time of chest pain
6. All subjects (male and female) must agree to use appropriate contraceptive methods (hormonal or barrier methods, abstinence) during study participation and up to 6 months of the last dosing, and women of childbearing age must test negative for pregnancy before dosing.

Exclusion Criteria:

1. Patients with a history of myocardial infarction who have received acute coronary thrombolysis, interventional therapy, or bypass surgery; A clear diagnosis of acute heart failure (Killip grade ≥III);
2. Severe arrhythmias that cannot be corrected;
3. Aortic dissection;
4. Severe liver and kidney dysfunction or severe consumption;
5. History of major surgery or hemorrhagic stroke within six months;
6. Previous history of malignant tumors;
7. Hypertensive patients with systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg after active antihypertensive treatment;
8. Clinically significant allergic reaction history, especially mannitol, drugs, protein preparations, biological products;
9. Patients who participated in other clinical studies within 3 months prior to screening;
10. Can not perform CMR examination;
11. Other conditions deemed unsuitable for inclusion by the investigators (for example, those whose coronary arteries other than the left anterior descending branch were judged by the investigators to require elective revascularization therapy at the same time or within 1 month).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage change of myocardial infarction area | Day 5、Day 90
  The percentage of myocardial infarction area was defined as the percentage of CMR delayed enhancement area in the entire left ventricular myocardium as measured by plane geometry of computer-assisted enhanced myocardium.Percentage change of myocardial infarction size =D5 percentage of myocardial infarction size -D90 percentage of myocardial infarction size

SECONDARY OUTCOMES:
Myocardial mass (g) | Day 5、Day 90
  Myocardial infarction area was defined as CMR delayed enhancement area, and myocardial mass (g) were calculated , and determined by plane geometry method of computer-aided enhanced myocardium. Myocardial infarction size change =D5 myocardial infarction size -D90 myocardial infarction size.
Myocardial volume (ml) | Day 5、Day 90
  Myocardial infarction area was defined as CMR delayed enhancement area, and volume (ml) were calculated, and determined by plane geometry method of computer-aided enhanced myocardium.Myocardial infarction size change =D5 myocardial infarction size -D90 myocardial infarction size.
Myocardial microvessel obstruction area change value | Day 5、Day 90
  Myocardial microvessel obstruction area change value =D5 microvessel obstruction area -D90 microvessel obstruction area
The change of CK-MB before and after administration | Before the first dose, 12 hours after the first dose, day 2, day 3, day 4
  CK-MB change value = CK-MB value before administration - CK-MB value after administration
The area under the CK-MB curve within 4 days | Before the first dose, 12 hours after the first dose, day 2, day 3, day 4
  CK-MB change value = CK-MB value before administration - CK-MB value after administration
Changes of left ventricular ejection fraction (LVEF) | Day 5、Day 90
  Left ventricular ejection fraction (LVEF) change =D90 LVEF-D5 LVEF
Changes of left ventricular end-systolic volume (LVESV) | Day 5、Day 90
  Left ventricular end-systolic volume (LVESV) change =D90 LVESV-D5 LVESV
Changes of left ventricular end-diastolic volume (LVEDV) | Day 5、Day 90
  Left ventricular end-diastolic volume (LVEDV) change = D90 LVEDV-D5 LVEDV

CONTACTS AND LOCATIONS:
Overall Officials: KeFei Dou, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No